CLINICAL TRIAL: NCT07224789
Title: Liquid Biopsy for Early Detection of Colorectal Cancer Using Circular RNA
Acronym: CIRCLE
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/CIRCLE
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: circRNA; Early cancer detection; non-coding RNA; CRC; liquid biopsy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Colorectal Cancer - Training Cohort: Patients with histologically confirmed colorectal adenocarcinoma (Stage I-III) enrolled in the training set. Plasma samples are collected before any surgery or therapy for cf-circRNA profiling.
  Interventions: Diagnostic Test: cf-circRNA assay
- Non-Disease Control - Training Cohort: Healthy individuals with no prior malignancy or major systemic disease, age- and sex-matched to the CRC group, included in the training set.
  Interventions: Diagnostic Test: cf-circRNA assay
- Colorectal Cancer - Validation Cohort: Independent cohort of patients with histologically confirmed colorectal adenocarcinoma (Stage I-III) from separate institutions, used to validate the diagnostic cf-circRNA signature. Plasma obtained prior to treatment.
  Interventions: Diagnostic Test: cf-circRNA assay
- Non-Disease Control - Validation Cohort: Independent cohort of healthy participants without malignant or inflammatory bowel disease, serving as external validation controls.
  Interventions: Diagnostic Test: cf-circRNA assay

INTERVENTIONS:
Diagnostic Test: cf-circRNA assay — Circular RNA detection in plasma or serum by RT-qPCR

SUMMARY:
Colorectal cancer (CRC) is a leading cause of cancer-related deaths worldwide. This study aims to develop a non-invasive liquid biopsy assay using plasma-derived cell-free circular RNAs (cf-circRNAs) for early and accurate detection of colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common malignancy and the second leading cause of cancer-related mortality worldwide. Despite the proven benefit of screening colonoscopy, its invasive nature, high cost, and low adherence rates limit its use for population-level early detection. Current non-invasive screening tools, such as fecal occult blood testing and stool DNA assays, offer limited sensitivity, particularly for early-stage or right-sided colorectal tumors.

Therefore, there is a growing clinical need for a highly sensitive, minimally invasive, and patient-compliant diagnostic approach that can complement existing screening modalities.

Circular RNAs (circRNAs) are a novel class of endogenous non-coding RNAs characterized by covalently closed loop structures formed through back-splicing. Unlike linear RNAs, circRNAs are resistant to exonuclease-mediated degradation and are remarkably stable in body fluids. They exhibit tissue- and cancer-specific expression patterns, suggesting strong potential as non-invasive biomarkers.

Emerging evidence demonstrates that cell-free circRNAs (cf-circRNAs) circulate in plasma or serum either freely or encapsulated within extracellular vesicles such as exosomes. These cf-circRNAs retain the molecular signatures of their tumor of origin and can be reliably quantified using reverse transcriptase-quantitative PCR (RT-qPCR) or next-generation sequencing (NGS)-based platforms.

The CIRCLED study (Circular RNA for Colorectal Cancer Detection) is designed as a multi-center, case-control, observational study aiming to (1) identify diagnostic circRNA candidates from RNA sequencing, and (2) validate a cf-circRNA diagnostic panel capable of differentiating CRC patients from healthy individuals and those with benign colorectal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Histologically confirmed colorectal cancer (Stage I-III)
* Availability of pre-treatment plasma samples
* Written informed consent provided

Exclusion Criteria:

* History of other active malignancies within the past 5 years
* Poor sample quality or hemolysis
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed colorectal adenocarcinoma (Stages I-III) Patients with benign colorectal diseases (adenoma, polyp) Healthy control individuals with no evidence of malignancy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  Proportion of early-stage (Stage I-II) colorectal cancer patients correctly identified as positive by the circRNA-based diagnostic model.

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  True Negative Rate: the probability of a negative test result, conditioned on the individual truly being negative
Proportion of correct predictions (true positives and true negatives) among the total cases (i.e., accuracy) | Through study completion, an average of 1 year
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data

REFERENCES:
- [Background] Dong Y, He D, Peng Z, Peng W, Shi W, Wang J, Li B, Zhang C, Duan C. Circular RNAs in cancer: an emerging key player. J Hematol Oncol. 2017 Jan 3;10(1):2. doi: 10.1186/s13045-016-0370-2. PMID 28049499
- [Background] Qu S, Yang X, Li X, Wang J, Gao Y, Shang R, Sun W, Dou K, Li H. Circular RNA: A new star of noncoding RNAs. Cancer Lett. 2015 Sep 1;365(2):141-8. doi: 10.1016/j.canlet.2015.06.003. Epub 2015 Jun 5. PMID 26052092
- [Background] Jeck WR, Sharpless NE. Detecting and characterizing circular RNAs. Nat Biotechnol. 2014 May;32(5):453-61. doi: 10.1038/nbt.2890. PMID 24811520
- [Background] Chen LY, Wang L, Ren YX, Pang Z, Liu Y, Sun XD, Tu J, Zhi Z, Qin Y, Sun LN, Li JM. The circular RNA circ-ERBIN promotes growth and metastasis of colorectal cancer by miR-125a-5p and miR-138-5p/4EBP-1 mediated cap-independent HIF-1alpha translation. Mol Cancer. 2020 Nov 23;19(1):164. doi: 10.1186/s12943-020-01272-9. PMID 33225938
- [Background] Xu H, Liu Y, Cheng P, Wang C, Liu Y, Zhou W, Xu Y, Ji G. CircRNA_0000392 promotes colorectal cancer progression through the miR-193a-5p/PIK3R3/AKT axis. J Exp Clin Cancer Res. 2020 Dec 14;39(1):283. doi: 10.1186/s13046-020-01799-1. PMID 33317596
- [Background] Long F, Lin Z, Li L, Ma M, Lu Z, Jing L, Li X, Lin C. Comprehensive landscape and future perspectives of circular RNAs in colorectal cancer. Mol Cancer. 2021 Feb 3;20(1):26. doi: 10.1186/s12943-021-01318-6. PMID 33536039
- [Background] Zhang Y, Luo J, Yang W, Ye WC. CircRNAs in colorectal cancer: potential biomarkers and therapeutic targets. Cell Death Dis. 2023 Jun 9;14(6):353. doi: 10.1038/s41419-023-05881-2. PMID 37296107
- [Background] Keum N, Giovannucci E. Global burden of colorectal cancer: emerging trends, risk factors and prevention strategies. Nat Rev Gastroenterol Hepatol. 2019 Dec;16(12):713-732. doi: 10.1038/s41575-019-0189-8. Epub 2019 Aug 27. PMID 31455888
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679